CLINICAL TRIAL: NCT03870984
Title: Efficacy of Walnuts and Hazelnuts on the Modification of the Lipid Content of Erythrocyte Membranes in Obese Children. A Randomised Controlled Trial.
Brief Title: Efficacy of Nuts in Obese Children.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Cristiano Fava, Professor, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VRINoci
Record Dates: First submitted 2019-03-06; First posted 2019-03-12 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Child Obesity
Keywords: obesity, children, nuts,
MeSH Terms: conditions — Pediatric Obesity; Obesity | interventions — Caloric Restriction; Nuts

STUDY DESIGN:
Intervention Model Description: Randomized design. Two arms in parallel with blinded operator.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- wNUTS, low-caloric diet plus nuts (Experimental): low-caloric diet personalized on single children's requirements plus nuts (15g hazelnuts+15g nuts without shell) for 3 months.
  Interventions: Dietary Supplement: wNUTS, low-caloric diet plus nuts; Other: w/oNUTS, low-caloric diet without nuts
- w/oNUTS, low-caloric diet without nuts (Other): low-caloric diet personalized on single children's requirements plus nuts (15g hazelnuts+15g nuts without shell) for 3 months.
  Interventions: Other: w/oNUTS, low-caloric diet without nuts

INTERVENTIONS:
Dietary Supplement: wNUTS, low-caloric diet plus nuts — 15g of nuts and 15g of hazelnuts in association with low caloric diet
  Arms: wNUTS, low-caloric diet plus nuts
Other: w/oNUTS, low-caloric diet without nuts — low caloric diet

SUMMARY:
Obesity is a problem of ever-growing importance, especially in industrialized countries, both in adults and in the pediatric population. Children and obese adolescents, like adults, have an increased risk, compared with normal-weight peers, to develop metabolic syndrome and atherosclerotic disease, pathophysiological basis of cardiovascular events. Alteration of the elastic properties of the arteries has been described previously in obese children and adolescents and is considered an initial marker of atherosclerotic vascular damage. The determination of the indices of arterial stiffness (PWV, Pulse Wave Velocity; AI, Augmentation Index, SI, Stiffness Index) is possible through techniques currently used for the determination of vascular function even in children.

Nuts and hazelnuts are rich in potentially beneficial substances including unsaturated fatty acids, especially omega-6 (present in both) and omega-3 (present only in nuts), Several clinical trials have already shown in adults a potential beneficial effect of the addition of different types of nuts (walnuts, hazelnuts, cashews, pistachios, etc.) on the characteristics of the metabolic syndrome also through their possible antioxidant effect and vasoactive. In children, some epidemiological studies have associated with a higher consumption of nuts reduced risk of hypertension, dyslipidemia, obesity and fasting glucose. The study will be conducted with a randomized design with two arms in parallel with blinded operator. The main objective of this study is to assess the efficacy of 15 grams of nuts and 15 grams of nuts a day in addition to a low calorie diet on the content of erythrocyte membranes of alpha-linolenic acid three months after the beginning of the trial in a group of obese children. Secondary objectives are to evaluate the efficacy of walnuts and hazelnuts in improving the systolic and/or diastolic blood pressure values, lipid profile, glucose and fasting insulin, vascular function.

DETAILED DESCRIPTION:
Obesity is a problem of ever-growing importance, especially in industrialized countries, widespread both in adults and in the pediatric population.

Children and obese adolescents, like adults, have an increased risk, compared with normal-weight peers, to develop high blood pressure, insulin resistance, diabetes, hyperlipidemia, fatty liver disease and the resulting long-term complications. This cluster of metabolic and hemodynamic risk factors, which is known as metabolic syndrome, greatly increases the risk of cardiovascular events in adults. Cardiovascular disease is the leading cause of mortality and morbidity in developed countries and are becoming even in developing countries. Atherosclerotic disease is the pathophysiological basis of cardiovascular events. Atherosclerosis is a multifactorial disease whose early stages of subclinical damage are documented much earlier in cardiovascular events with non-invasive tests. The determination of the indices of arterial stiffness (PWV, Pulse Wave Velocity; AI, Augmentation Index, SI, Stiffness Index) is possible through techniques currently used for the determination of vascular function even in children. The alteration of the elastic properties of the arteries has been described previously in obese children and adolescents and is considered initial marker atherosclerotic vascular damage. Fats particularly saturated fats, without adequate intake of polyunsaturated fat, may facilitate the development of obesity.

The consumption of some specific foods including dried fruit (in a broad sense including walnuts, hazelnuts, almonds, cashews, etc.) within a reduced calorie diet is considered to be a promising approach in the prevention and care of the different components of the metabolic syndrome. The nuts and hazelnuts are rich in potentially beneficial substances including unsaturated fatty acids, especially omega-6 (present in both) and omega-3 (present only in nuts), L-arginine, fiber, minerals, vitamin E, fitosetrols and polyphenols.

Several clinical trials have already shown in adults a potential beneficial effect of the addition of different types of nuts (walnuts, hazelnuts, cashews, pistachios, etc.) on the characteristics of the metabolic syndrome also through their possible antioxidant and vasoactive effect .

In children, some epidemiological studies have associated a higher consumption of nuts with reduced risk of hypertension, dyslipidemia, obesity and fasting glucose alteration.

Our group conducted a study in obese children observing an inverse relationship between omega-6 polyunsaturated fatty acids, contained in large amounts in walnuts, and certain features of metabolic syndrome, such as waist circumference, triglycerides, fasting insulin, systolic blood pressure of 24-hours, suggesting a possible beneficial effect. The project was financed by health ministry and included also the present Protocol ("Obesity, hypertension and subclinical vascular damage in children: the role of dietary factors and lipid mediators. An epidemiological and translational study. "Project Code: GR-2011-02349630).

From arachidonic acid, the main omega-6 type polyunsaturated fatty acids (PUFA), certain metabolites are produced via cytochrome P450 which have vasoactive and natriuretic effect: 20-Hydroxyeicosatetraenoic acid (20-HETE), the epoxyeicosatrienoic acids (EETs) and dihydroxyeicosatrienoic acids (DHETs). From numerous studies in animal models and some human studies, it is known that these metabolites via cytochrome P450 may be involved both in the homeostasis of blood pressure pressure and in the development of hypertension. In particular, plasmatic 20-HETE has a vasoconstrictor effect while EETs are vasodilators; both exert renal natriuretic effect. Our study intends to verify if in a group of obese children, a low-calorie diet that contains a portion of walnuts and hazelnuts, can change the content of polyunsaturated fatty acids in erythrocyte membranes, particularly alpha-linolenic acid. This could result in possible beneficial effects on the characteristics of the metabolic syndrome in obese children, like an improvement of waist circumference, blood pressure, HDL cholesterol, triglycerides and blood sugar. Our study also intends to acquire information on the effect of the addition of walnuts and hazelnuts and the metabolites of polyunsaturated fatty acids omega-3 and omega-6 metabolized by cytochrome P450 that derives from these nuts in change vessel elasticity.

2. STUDY DESIGN The study will be conducted with a randomized design (two arms in parallel with blinded operator). Doctors in charge of vascular measurements and laboratory technicians will not know which of the two groups analyzed will only have taken the low-calorie diet and who will have assumed the low-calorie diet with walnuts and hazelnuts.

3. PURPOSE OF THE STUDY

The main objective of this study is to assess the efficacy of 15 grams of nuts and 15 grams of nuts a day in addition to a low calorie diet, in modifying the content of of alpha-linolenic acid in erythrocyte membranes evalutated three months after the beginning of the assumption in a group of obese children.

Secondary objectives are:

To evaluate the efficacy of walnuts and hazelnuts in improving in obese children:

* the systolic and/or diastolic blood pressure values;
* metabolic disorders (in particular of the lipid profile: LDL, HDL, triglycerides, and glucose: glucose and fasting insulin);
* vascular function measured by tonometry (PWV and PWA), and ultrasonography (carotid distensibility).
* the modifications of the profile of eicosanoids via CYP450 in plasma and urine

To evaluate:

- the relationship between intake of nuts and hazelnuts, fatty acid profile of erythrocyte membranes and eicosanoids via CYP450, the components of the metabolic syndrome including the blood pressure and vascular elasticity.

ELIGIBILITY:
Inclusion Criteria:

* obese subjects (BMI ≥ 95th percentile for age and sex; reference tables for WHO BMI);
* Aged between 6 and 17 years;
* Signature applied in the informed consent by both parents and consent of the child

Exclusion Criteria:

* chronic liver diseases (hepatitis, cirrhosis).
* Chronic renal failure (serum creatinine> 1.2 mg / dL).
* Malignancies.
* Diabetes (fasting blood glucose ≥ 126 mg / dl or therapy with oral hypoglycemic drugs or insulin).
* cholesterol-lowering or antihypertensive terapy.
* Notes allergies to nuts or hazelnuts or food intolerance to nuts and/or hazelnuts.
* Treatment of less than 6 weeks with any medication which can interfere with fecal microbiota (particularly antibiotics or laxatives).

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
ALA change | baseline compared to post-treatment (ie, after 3 months of treatment)
  Primary outcome is to compare percentage of fatty acids in erythrocyte membranes (in particular alpha-linolenic acid, ALA) with the content of other membrane-bound fatty acids. It will be compared in the two groups the ALA delta (delta%) between measurement at baseline compared to post-treatment (ie, after 3 months of treatment).

SECONDARY OUTCOMES:
LA change | baseline compared to post-treatment (ie, after 3 months of treatment)
  to compare percentage of fatty acids in erythrocyte membranes (in particular linoleic acid, LA) with the content of other membrane-bound fatty acids. It will be compared in the two groups the ALA delta (delta%) between measurement at baseline compared to post-treatment (ie, after 3 months of treatment).
ABPM change | baseline compared to post-treatment (ie, after 3 months of treatment)
  To compare ambulatory blood pressure (mmHg) measured by validated devices (A&D TM-2430; in the week preceding the beginning of the assumption of diet plus or minus nuts/hazelnuts) and after 3 months from randomization in the two arms.
OFFICE BLOOD PRESSURE change | baseline compared to post-treatment (ie, after 3 months of treatment)
  To compare mean arterial pressure obtained during the medical examination (mmHg) by oscillometric validated device in children (Omron 705 IT; average of three measurements) prior to randomization and after 3 months of diet intake plus or minus nuts/hazelnuts.
HDL-cholesterol change | baseline compared to post-treatment (ie, after 3 months of treatment)
  To compare HDL-cholesterol
triglycerides change | baseline compared to post-treatment (ie, after 3 months of treatment)
  To compare triglycerides
glucose change | baseline compared to post-treatment (ie, after 3 months of treatment)
  To compare plasma glucose
WAIST CIRCUMFERENCE change | baseline compared to post-treatment (ie, after 3 months of treatment)
  To compare waist circumference change in the 2 arms prior to randomization and after 3 months of diet intake plus or minus nuts/hazelnuts.
WEIGHT change | baseline compared to post-treatment (ie, after 3 months of treatment)
  To compare weight change in the 2 arms prior to randomization and after 3 months of diet intake plus or minus nuts/hazelnuts.
PWA (Augmentation Index; AIx) change | baseline compared to post-treatment (ie, after 3 months of treatment)
  To compare AIx change as measured by pulse wave analysis (PWA) by SphygmoCor XCEL and in the 2 arms prior to randomization and after 3 months of diet intake plus or minus nuts/hazelnuts.
cfPWV change | baseline compared to post-treatment (ie, after 3 months of treatment)
  To compare carotid femoral pulse wave velocity (PWV) change measured by tonometer (SphygmoCor XCEL) in the 2 arms prior to randomization and after 3 months of diet intake plus or minus nuts/hazelnuts.
carotid distensibility (cDC) change | baseline compared to post-treatment (ie, after 3 months of treatment)
  To compare cDC change measured by ultrasound in the 2 arms prior to randomization and after 3 months of diet intake plus or minus nuts/hazelnuts.
plasma EETs change | baseline compared to post-treatment (ie, after 3 months of treatment)
  To compare plasma epoxyeicosatrienoic acids, metabolites of arachidonic acid vis CYP450
plasma DHETs change | baseline compared to post-treatment (ie, after 3 months of treatment)
  To compare plasma dihydroxyeicosatrienoic acids, metabolites of EETs via sEH
urine DHETs change | baseline compared to post-treatment (ie, after 3 months of treatment)
  To compare urine dihydroxyeicosatrienoic acids, metabolites of EETs via sEH
plasma 20-HETE change | baseline compared to post-treatment (ie, after 3 months of treatment)
  To compare plasma 20-hydroxyeicosatetraenoic acids, metabolites of arachidonic acid via CYP450
urine 20-HETE change | baseline compared to post-treatment (ie, after 3 months of treatment)
  To compare urine 20-hydroxyeicosatetraenoic acids, metabolites of arachidonic acid via CYP450
plasma EEQs change | baseline compared to post-treatment (ie, after 3 months of treatment)
  To compare plasma epoxyeicosatetraenoic acids, metabolites of eicosapentaenoic acid via CYP450
plasma EDPs change | baseline compared to post-treatment (ie, after 3 months of treatment)
  To compare plasma epoxydocosapentaenoic acids, metabolites of docosahexaenoic acid via CYP450
MICROBIOTA change | baseline compared to post-treatment (ie, after 3 months of treatment)
  To compare profile of the faecal microbiota by metagenomic of the gene sequences coding for the 16S rRNA prior to randomization and after 3 months of diet intake plus or minus nuts/hazelnuts.

CONTACTS AND LOCATIONS:
Overall Officials: Cristiano Fava, professor, Principal Investigator — Universita di Verona
Locations (1):
- AOUI Verona, Verona, VR, Italy